CLINICAL TRIAL: NCT01605513
Title: Phase I Clinical Trial of PEG-IFN-SA in HCV Disease: Evidence for Drug Safety, Tolerance, and Antiviral Activity
Brief Title: Safety Study of Recombinant Interferon Variant(PEG-IFN-SA) to Treat HCV Disease
Acronym: PEG-IFN-SA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yanhua Ding, associate professor, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011L0901
Record Dates: First submitted 2012-05-10; First posted 2012-05-25 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C Virus
Keywords: recombinant interferon, tolerated, effective
MeSH Terms: conditions — Hepatitis C | interventions — Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- recombinant interferon (Experimental): PEG-IFN-SA 1.0μg/kg for 12 times, Peginterferon alfa-2a 180 μg for 12 times, PEG-IFN-SA 1.5 μg/kg for 12 times, PEG-IFN-SA 2 μg/kg for 12 times, PEG-IFN-SA 3 μg/kg for 12 times, PEG-IFN-SA 1.5μg/kg + ribavirin 0.45g/bid group for 12 times, Intergen 15μg/48hours for 7 times, ribavirin 0.45g/bid for 10 times
  Interventions: Drug: interferon

INTERVENTIONS:
Drug: interferon — PEG-IFN-SA (new interferon) was injected subcutaneously one times per week for 12 times.

SUMMARY:
The purpose of this study is to determine whether PEG-IFN-SA is safe, tolerant and effective in the treatment of HCV patients.

DETAILED DESCRIPTION:
Chronic infection with the hepatitis C virus (HCV) is a significant public health problem in china. Progressive liver disease, as a result of chronic HCV infection, usually develops slowly over 20-50 years and may lead to cirrhosis, hepatocellular carcinoma, liver failure and eventual death. Symptoms are typically mild and non-specific but nevertheless can cause a decrease in quality of life. Peginterferon alfa and ribavirin combination therapy is currently used in the china for treatment of chronic HCV. Successful treatment is considered to be attainment of a sustained virological response (SVR), defined as undetectable serum HCV ribonucleic acid (RNA) 6 months after cessation of treatment.

PEG-IFN-SA is a new recombinant interferon variant. Its N-terminus is modified by 20KD molecular weight single-methoxy polyethylene glycol (PEG). It consists of 171 amino acids before modification. PEG-IFN-SA is reorganization, unnatural existence and a new type of interferon (171Arg126Asp171IFN) after modification. The safety, tolerance and antiviral activity of PEG-IFN-SA was tested in adults with HCV infection.

PEG-IFN-SA was injected subcutaneously one times per week for 12 times. Peginterferon alfa-2a (Pegasys) is the positive control drug. 80 patients were randomly assigned to eight groups (PEG-IFN-SA 1.0μg/kg, Peginterferon alfa-2a 180 μg, PEG-IFN-SA 1.5 μg/kg，PEG-IFN-SA 2 μg/kg， PEG-IFN-SA 3 μg/kg，PEG-IFN-SA 1.5μg/kg + ribavirin 0.45g/bid group，Intergen 15μg/48hours for 7 times and ribavirin 0.45g/bid for 10 times).

Clinical and biological adverse effects were recorded every week such as headache, nausea and vomiting. HCV RNA level was tested by COBAS Taqman HCV Test system of Roche. Blood cell counts were tested using an automatic cell counter such as WBC, neutrophil, PLT and HGB. Biochemical indicators were tested by automatic biochemical analysis instrument.

ELIGIBILITY:
Inclusion Criteria:

1. enrolled voluntarily, can understand and sign informed consent;
2. More than 18 years and less than 65 years;
3. body mass index (BMI) is at 18 - 26;
4. anti-HCV antibodies and / or HCV RNA positive, and / or other evidence of chronic hepatitis C;
5. HCV RNA level ≥ 2000IU/ml (or equal to this viral load);
6. Women's urine pregnancy test was negative, and the subjects (male subjects) is willing to have no pregnancy plans at next 18 months. (7) ALT is within 6 times of the upper limit of normal

Exclusion Criteria:

1. pregnant women, lactating women or plan to pregnant the next 18 months.
2. mental disorder, including history of mental illness (especially the history of depression or depressive tendencies, epilepsy, etc.);
3. The patient who received interferon therapy within the past six months or had no response at previous interferon therapy.
4. The patient who used a strong immune regulator over two weeks with three months before screening, such as adrenocorticotropic hormone, thymosin of α1, thymus 5 peptide.
5. The patient who used hepatotoxic drugs with 6 months before screening, such as dapsone, erythromycin, fluconazole, ketoconazole, rifampin.
6. co-infection with other viruses (HAV, HBV, HEV, the HIV, EBV, CMV) .
7. patients with a history of hepatocellular carcinoma (HCC), or may had hepatocellular carcinoma evidence, such as imaging of suspicious nodules, or AFP abnormal (AFP> 200ng/mL). FibroScan value greater than or equal to F3 at Screening
8. other causes of liver disease: a chronic alcoholic hepatitis, drug-induced hepatitis, autoimmune liver disease, nonalcoholic steatohepatitis.
9. autoimmune diseases, including psoriasis, systemic lupus erythematosus, thrombocytopenic purpura, and so on.
10. heart and vascular system diseases, a history of myocarditis, hypertension, coronary heart disease, pathological arrhythmia, stroke.
11. endocrine system diseases, including thyroid disease, diabetes, etc.
12. pulmonary diseases, including invasive pulmonary disease, pneumonia, shortness of breath.
13. Eye diseases, including retinopathy, retinopathy.
14. chronic infectious disease history (history of tuberculosis).
15. chronic kidney disease, serum creatinine level> 1.5 times upper limit of normal at screening, renal insufficiency, renal anemia history.
16. anemia (including thalassemia, sickle hemoglobin, anemia), and hemophilia.
17. peptic ulcer not controlled, colitis, pancreatitis and others.
18. malignancies.
19. peripheral blood checking: white blood cell count <3 × 109 / L; neutrophil count <1.5 x 109 / L; platelet count <90 × 109 / L; hemoglobin was less than the normal reference limit.
20. serum total bilirubin> 2 times normal maximum reference value (ULN); serum albumin <35g / L; a history of decompensated cirrhosis evidence.
21. evidence of drug addiction (including excessive alcohol intake, average alcohol consumption: men> 40g / day; women> 20g / day, equivalent to 50 degrees white wine 100ml / day and 50ml / day) within one year before screening.
22. a serious history of drug and food allergy, especially towards the test drug (interferon, ribavirin).
23. plans to accept an organ transplant or have organ transplant.
24. participated other clinical trials before 3 months at screening
25. The researchers judged the patients have other factors which may influence the experiment.

ribavirin exclusion criteria:

1. women Hgb <12g/dl or men Hgb <13gdl at screening.
2. anemia patients (eg, thalassemia, spherocytosis hyperlipidemia, gastrointestinal bleeding history) or suspected anemia patients.
3. patients have a history of coronary artery disease or patients with cerebrovascular disease should not join this study, hemoglobin decline up to 4g/dl (it may be observed in the ribavirin treatment).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The proportions of absence of detectable HCV RNA after the 12th treatment | 12th week

SECONDARY OUTCOMES:
The proportions of absence of detectable HCV RNA after the 4th and 8th treatment | 4th and 8th week
HCV RNA levels after the 4th, 8th and 12th treatment | the 4th, 8th and 12th week
The test of Liver function | the 2th, 4th, 6th, 8th,10th and 12th week
  Liver function test:TBIL,IBIL, ALT, AST;
The test of Kidney function | the 2th, 4th, 6th, 8th,10th and 12th week
  Kidney function test:BUN, CR;
The test of Peripheral blood | the 2th, 4th, 6th, 8th,10th and 12th week
  Peripheral blood detection:WBC, RBC, HgB,PLT, neutrophil

CONTACTS AND LOCATIONS:
Overall Officials: yanhua ding, associate professor, Study Director — First Hospital, Jilin University
Locations (1):
- Phase One Clinical Trial ward, First Hospital, Jilin University, Changchun, Jilin, China